CLINICAL TRIAL: NCT00061282
Title: Clotrimazole Enemas for Pouchitis in Children and Adults
Acronym: CAPTURE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding Horizon
Sponsor: Web (Other)
Responsible Party: Sponsor-Investigator, Web, Assistant Professor of Pediatrics, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2202
Record Dates: First submitted 2003-05-23; First posted 2003-05-26 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Ulcerative Colitis; Pouchitis; Ileitis; Inflammatory Bowel Disease
Keywords: Pouchitis; Colitis; Ileitis
MeSH Terms: conditions — Colitis, Ulcerative; Pouchitis; Ileitis; Inflammatory Bowel Diseases; Colitis | interventions — Clotrimazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: Clotrimazole
- 2 (Active Comparator): Clotrimazole Therapy
  Interventions: Drug: Clotrimazole
- 3 (Active Comparator): Clotrimazole Therapy
  Interventions: Drug: Clotrimazole

INTERVENTIONS:
Drug: Clotrimazole — One retention enema, administered nightly

SUMMARY:
Colectomy with creation of an ileal pouch (IPAA) is now the treatment of choice for patients with ulcerative colitis that is resistant to existing medical therapies. The development of inflammation in these ileal reservoirs, a clinical entity referred to as pouchitis, is the most common long-term complication of this procedure and can affect 50-60% of adults and children. We have previously demonstrated that clotrimazole (delivered as a rectal suppository) is generally safe, effective, and displays poor systemic absorption when used in pediatric and adults with active pouchitis. We saw clinical benefit in patients with pouch disease that had previously failed to respond to standard antibiotic, steroid, or immunosuppressive therapies. The clinical trial outlined here will define the effectiveness and safety of topical clotrimazole therapy (delivered as a rectal enema) in pediatric (aged greater than two years) and adult patients with pouchitis.

Subjects in this study will be randomly assigned to receive either placebo (no active drug, 4 subjects) or one of two clotrimazole therapy groups: 2500 mg/day (8 subjects) or 4000mg/day (8 subjects). No washout period is required, and subjects will be allowed to continue their existing anti-inflammatory medications during their participation in the study. Clotrimazole will be delivered nightly in the form of an enema. Subjects will undergo flexible sigmoidoscopy (pouchoscopy) prior to and again after completing one month of study therapy, and pouch disease activity will be graded at after each procedure using the Pouchitis Disease Activity Index (PDAI). Clinical improvement will be defined as a drop in PDAI score. If the drop in PDAI scores between placebo and either active clotrimazole treatment group is not significant, and no subject experiences what are determined to be study-related adverse effects, a second cohort of subjects will be recruited and studied after receiving one month of either placebo (4 subjects), 6000 mg/day clotrimazole (8 subjects), or 7500mg/day clotrimazole (8 subjects).

Subjects will be assessed for adverse effects at the midpoint of the study. Clotrimazole blood levels will be measured during the first and last day of study participation. In addition, adults will complete a health related quality of life assessment at baseline and after completing study drug therapy.

All subjects will be eligible for one month of open-label study drug therapy after completing one month of study drug therapy.

ELIGIBILITY:
* Age greater than 2 years
* Availability of Parent or Legal Guardian (for those less than 2 years of age).
* History of ulcerative colitis treated with colectomy and ileal pouch
* Diagnosis of acute or chronic pouchitis

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2002-09-30 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Improvement in Pouchitis Disease Activity Index (PDAI) | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Rufo, MD, MMSc, Principal Investigator — Children's Hospital and Harvard Medical School
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Crohn's and Colitis Foundation of America — http://ccfa.org